CLINICAL TRIAL: NCT06855251
Title: SENSing Inner BodiLy State: Understanding the Role of Interoception in obEsity
Acronym: SENSIBLE
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C404
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Body Representation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Right-handed women diagnosed with obesity are consecutively recruited during their rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders are exclusion criteria.
  Interventions: Behavioral: The crossmodal dual-task
- Controls: Age-matched, right-handed, healthy women (i.e., with no history of eating disorders) are recruited outside the hospital through personal contacts of the researchers and word-of-mouth.
  Interventions: Behavioral: The crossmodal dual-task

INTERVENTIONS:
Behavioral: The crossmodal dual-task — Two main sensory tasks performed together:
  1. the visual task, in which participants are requested to monitor visual stimuli presented on a computer screen and to detect the "deviant" target" as soon as possible. The target changes across blocks: in half of the trials, participants will have to respond to food stimuli presented together with irrelevant non-food stimuli (food target condition); in the other half conditions, participants will have to respond to non-food stimuli presented together with irrelevant food stimuli (non-food target condition). For each participant, we will collect the Reaction Time in milliseconds only for the valid responses, and the level of Accuracy in percentage.
  2) The interoceptive task, in which participants are requested to monitor their heartbeat presented through headphones and registered through pulse oximetry. Participants will judge the level of asynchrony between their heartbeat and the auditory cue.

SUMMARY:
Successfully perceiving the flow of interoceptive cues and integrating them with exteroceptive information are fundamental aspects of countering the body's inherent instability and guaranteeing homeostatic regulation. This process deeply affects cognitive/emotional functioning and general health. Recently, it has been suggested that an important signature underpinning obesity might be an interoceptive dysfunction in perceiving internal body signals and/or integrating them with information from the external environment. There is evidence that interoceptive deficits correlate with Body Mass Index (BMI), but it is still largely unclear how different measures and facets of interoception are related to high BMI and eating behaviour. Within this framework, it is mandatory to understand the role of interoception in obesity at perceptual, cognitive, and emotional levels. One open issue regards the relationships between interoceptive signals and the reactivity to external food cues.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed individuals diagnosed with obesity
* In rehabilitative treatment at the Istituto Auxologico

Exclusion Criteria:

* Concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with obesity were consecutively recruited during their rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual detection velocity | At the moment of the experiment
  Reaction Time in milliseconds only for the valid responses in the visual task
Interoceptive judgement | At the moment of the experiment
  Individual's judgement from 0 (no synchronicity) to 100 (maximum synchronicity) between between the auditory stimulus and own heartbeat in the heartbeat detection task

SECONDARY OUTCOMES:
Visual detection accuracy | At the moment of the experiment
  Percentage of the correct answers in the "No-Go" trials in the visual task.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Scarpina, PhD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy